CLINICAL TRIAL: NCT03954795
Title: The Comparison of Analgesic Sparing Effects of Oblique Subcostal Transversus Abdominis Plane Block (OSTAP) and Transversus Abdominis Plane Block (TAP) in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: OSTAP Versus TAP for Postoperative Pain Management in Laparoscopic Cholecystectomy Patients
Acronym: OSTAP/TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, associated professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BAUA
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Pain Postoperative
Keywords: TAP OSTAP Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: TAP Block (Active Comparator): TAP Block performed from the petit triangle ( anterior axillary line and iliac crest.)
  Interventions: Procedure: TAP
- Group 2: OSTAP Block (Active Comparator): Modified TAP (OSTAP) block performed from the medial of linea semilunaris applying local anesthetic to the area between xiphoid and anterior iliac crest.
  Interventions: Procedure: OSTAP
- No Block (No Intervention): No interventions

INTERVENTIONS:
Procedure: TAP — Classic TAP block performed through the petit triangle (the anterior axillary line and iliac crest)
  Arms: Group 1: TAP Block
Procedure: OSTAP — Modified TAP (OSTAP) block performed from the medial of linea semilunaris applying local anesthetic to the area between xiphoid and anterior iliac crest.
  Arms: Group 2: OSTAP Block

SUMMARY:
The aim of the study is to compare the effectiveness and opioid sparing effects of TAP and OSTAP in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic cholecystectomy were separated into 3 groups. Group 1: Received TAP block Group 2: Received OSTAP Group 3: No Block Standard General Anesthesia was induced and maintained in all patients. At the end of the operation patient controlled analgesia with morphine was applied to all patients.

Pain scores were evaluated at 0,2,4,6,12,24 hours postoperatively. Total morphine consumption and pain scores were compared.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic cholecystectomy
* ASA status I-II

Exclusion Criteria:

* Local anesthetic allergy
* Coagulopathy
* Infection at procedure site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain scores throughout time evaluated by VAS | Pain scores will be recorded for 24 hours postoperatively. The first measure will be taken immediately after surgery (time 0) and then at 2. 4. 6. 12. 24. hours.
  Pain scores are going to be evaluated via VAS score. The VAS score will be scored between 0-10. 0 points is defined as no pain and 10 points is the most severe pain imaginable by the patient. A higher VAS score reflects a poor pain control.
Change in opioid Sparing effect measured through morphine amount delivered by a patient controlled analgesia device. | The amount of Morphine demanded by the patient will be recorded for 24 hours postoperatively. The first measure will be taken immediately after surgery (time 0) and then at 2. 4. 6. 12. 24. hours.
  The amount of morphine demand of the patient measured through morphine delivery by the patient controlled analgesia device
Amount of total intraoperative remifentanil infusion | At the end of surgery.
  The total amount of infused remifentanil throughout the surgery will be recorded from the infusion device.